CLINICAL TRIAL: NCT06824402
Title: A Prospective, Randomized Clinical Trial to Evaluate the Feasibility of Miniature Cryoprobe Biopsy to Detect Acute and Chronic Lung Transplant Rejection in Lung Transplant Recipients
Brief Title: Cryoprobe Biopsy and Chronic Rejection in Lung Transplant Recipients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, John O. Joerns, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 23-011339
Record Dates: First submitted 2025-02-07; First posted 2025-02-13 (Actual); Last update posted 2025-04-21 (Actual); Status verified 2025-04

CONDITIONS: Lung Transplant Rejection
Keywords: Lung Transplant; Bronchoscopy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Allocation will not be known to either the patient or bronchoscopist until the intra-procedural randomization timepoint, after which blinding of the bronchoscopist is not possible due to the nature of the procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Cryoprobe Biopsy Method (Experimental): Cryoprobes which are flexible catheters that can be passed through the channel of a bronchoscope. Rapid cooling of tissue results from the Joule-Thomson effect which causes tissue to freeze and adhere to the probe. The biopsy is obtained by subsequently avulsing small fragments of tissue.
  Interventions: Device: Cryoprobe Biopsy
- Forceps Biopsy Method (Active Comparator): Olympus disposable EndoJaw is used to obtain samples as per the standard of clinical care usually resulting in crush artifact.
  Interventions: Device: Forceps Biopsy

INTERVENTIONS:
Device: Forceps Biopsy — 10-12 transbronchial lung biopsies will be obtained using standard of care biopsy forceps: Olympus disposable EndoJaw (FB-211), Olympus, USA
  Arms: Forceps Biopsy Method
Device: Cryoprobe Biopsy — 3 transbronchial lung biopsies of two separate lobes will be obtained using a flexible cryoprobe: single-use, ø 1.1 mm (Erbe Elektromedizin GmbH, 20402-401) used with ERBECRYO 2 (Erbe Elektromedizin GmbH, 10402-000
  Arms: Cryoprobe Biopsy Method

SUMMARY:
The goal of this clinical trial is to evaluate which biopsy collection method helps to better diagnose rejection and relevant pathologic findings in lung transplant recipients. The main questions it aims to answer are:

Does the 1.1 mm cryoprobe or the biopsy forceps provide better quality samples of lung tissue for detecting rejection in transplant recipients?

How much tissue is adequate for lung transplant 1.1 mm cryobiopsy samples as compared to biopsy forceps?

Which samples received by the pathologist did they find they were most confident to exclude rejection, based on their satisfaction with the samples?

Which collection method has the least amount of procedural time?

Researchers will compare lung tissue samples obtained using a 1.1mm cryoprobe and a biopsy forceps during the lung transplant.

Participants will:

Be randomly assigned to receive either the cryoprobe or biopsy forceps collection method at the time of biopsy.

Assessed for any adverse events following the biopsy for up to 30 days after transplant.

DETAILED DESCRIPTION:
The purpose of this 1:1 randomized clinical trial is to compare the histological quality and diagnostic yield of tissue samples acquired using a 1.1 mm cryoprobe with those obtained with biopsy forceps in lung transplant recipients for graft surveillance.

ELIGIBILITY:
Inclusion Criteria

* Male and female lung transplant recipients age >18 at the time of informed consent
* Patients clinically meet indication for post-transplant lung biopsy or planned routine surveillance and have been scheduled for bronchoscopy with transbronchial biopsy.
* Be willing and able to sign the informed consent.

Exclusion Criteria

* Patients with known bleeding diathesis
* Platelet count <50,000 per μL within 14 days of the biopsy procedure
* Current use of systemic anticoagulation or antiplatelet therapy without the ability to hold therapy for the recommended amount of time prior to an invasive procedure (aspirin monotherapy is acceptable)
* Inability or unwillingness to give informed consent or study procedures
* Pregnant or nursing females, or females who intend to become pregnant
* Females of child-bearing potential who decline a pregnancy test prior to enrollment
* If an investigator does not feel that this study is in the subject's best interest or would be a good fit for the study.
* International Normalized Ratio (INR) >1.5
* Do Not Resuscitate (DNR) status
* Do Not Intubate (DNI) status
* Single lung transplant recipients

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Quality and diagnostic yield of tissue samples | Baseline
  Histological accessibility grade is determined by the pathologist according to the Lung Allograft Standard Histological Analysis (LASHA) scale and the 2007 Revision of the 1996 working formulation for the Standardization of Nomenclature in the Diagnosis of Lung Rejection, published by the ISHLT.

SECONDARY OUTCOMES:
Time duration | Baseline
  Duration of each individual biopsy procedure from insertion of the bronchoscope after airway has been secured until bronchoscope is withdrawn. .
Tissue sample adequacy | Baseline
  Number of biopsy samples that are adequate to determine rejection based on the presence of well expanded alveoli, as determined by the pathologist.

CONTACTS AND LOCATIONS:
Overall Officials: John Joerns, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No